CLINICAL TRIAL: NCT04781998
Title: Is Pharmacological Treatment With the Glucagon-like Peptide-1 Receptor Agonist Liraglutide 3mg (Saxenda®) Once-daily a Viable Treatment for Weight Management in Forensic Psychiatry Patients? A Feasibility Study.
Brief Title: Is Saxenda® a Viable Treatment of Obese Patients in Forensic Psychiatry?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SaxPsychiatry
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Mental Disorder; Metabolic Disturbance; Feasibility; Overweight and Obesity; Liraglutide
MeSH Terms: conditions — Mental Disorders; Overweight; Obesity | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: An open-label, multi-centre, 26-weeks clinical feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- liraglutide 3 mg (Saxenda®) once-daily (Experimental)
  Interventions: Drug: liraglutide 3 mg (Saxenda®) once-daily

INTERVENTIONS:
Drug: liraglutide 3 mg (Saxenda®) once-daily — Liraglutide 3 mg (Saxenda®) 6 mg/ml, 3 ml pre-filled pen-injector. The injection is administered subcutaneously. The initial daily dose will be 0.6 mg liraglutide (Saxenda®) for one week. If tolerated patients increase the dose by +0.6 mg each week until the full maintenance of 3 mg is reached (week 1: 0.6 mg, week 2: 1.2 mg, week 3: 1.8 mg, week 4: 2.4 mg, week 5-26: 3.0 mg. If necessary, a longer titration period is accepted). If the lowest tolerated dose is less than 1.8 mg of liraglutide (Saxenda®) once-daily after 12 weeks from inclusion, the patient will be excluded from the study.

SUMMARY:
An open-label, multi-centre, 26-weeks clinical feasibility study. The objective is to explore whether Saxenda could be a feasible choice in the treatment of overweight, obesity and weight-related medical problems, in patients diagnosed with a severe mental illness and hospitalized at a forensic department in Denmark. We wish to determine the viability of the daily Saxenda®-injection treatment in this specific patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Informed oral and written consent
2. Diagnosed with a mental illness according to the criteria of ICD10
3. Hospitalised at a forensic psychiatric department during the full inclusion period
4. Age 18 years to 65 years (both included)
5. BMI ≥27 kg/m2 with one or more weight-related comorbidities (sleep apnea, hypertension (BT ≥ 140/90 mmHg with no antihypertensive treatment. BT ≥ 130/80 mmHg with antihypertensive treatment), dyslipidaemia (LDL cholesterol ≥ 3 mmol/L), pre-diabetes (HbA1c 39-47 mmol/mol) or type 2 diabetes (HbA1c ≥ 48 mmol/mol)) or BMI ≥30 kg/m2

Exclusion Criteria:

1. Any use of coercive measures according to the Danish law for Mental Health/Psykiatriloven (as defined in "Informationsbekendtgørelsen § 10").
2. Fertile females of child-bearing potential who are pregnant, breast-feeding or have the intention of becoming pregnant
3. Women who are not willing to use an adequate contraceptive considered as highly effective (IUD or hormonal contraception during the full length of the study
4. Impaired hepatic function (plasma liver transaminases >2 times the upper normal limit)
5. Impaired renal function (serum creatinine >150 μmol/l and/or macroalbuminuria)
6. Impaired pancreatic function (acute or chronic pancreatitis and/or plasma amylase >2 times the upper normal limit)
7. Cardiac problems defined as decompensated heart failure (NYHA class III/IV), unstable angina pectoris and/or myocardial infarction within the last 12 months
8. Hypertension with systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg
9. Any condition that the investigator feels would interfere with trial participation
10. Use of weight-lowering pharmacotherapy within the preceding 3 months
11. Type 1 diabetes
12. Patients treated with insulin
13. Patients treated with other GLP-1 receptor agonist medicines
14. Known allergy to liraglutide or any of the ingredients in Saxenda®

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the number of "completers" | 26 weeks
  Feasibility in this study is defined as a minimum of 75% completers with a confidence interval of ±10%.

SECONDARY OUTCOMES:
Reason(s) for drop-out | 26 weeks
  The reason for withdrawal may be the withdrawal of consent, any use of coercive measures, failure to maintain a present level of compliance with the clinical trial medication
Changes in body weight | 26 weeks
  Kg
HbA1c | 26 weeks
  mmol/mol
blood pressure | 26 weeks
  mmHg
heart rate | 26 weeks
  Beats/minute
FIB-4 score | 26 weeks
  index
lipid profile | 26 weeks
  mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Centre Sct.Hans. Forensic Mental Health Services in the Capitol Region of Denmark., Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No